CLINICAL TRIAL: NCT02244125
Title: A Multicenter Open Label Phase II Study of Pomalidomide and Cyclophosphamide and Dexamethasone in Relapse/Refractory Multiple Myeloma Patients Who Were First Treated Within the IFM/DFCI 2009 Trial
Brief Title: A Multicenter Open Label Phase II Study of Pomalidomide and Cyclophosphamide and Dexamethasone in Relapse/Refractory Multiple Myeloma Patients Who Were First Treated Within the IFM/DFCI 2009 Trial (PCD)
Acronym: PCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Intergroupe Francophone du Myelome (Network); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2013-05
Record Dates: First submitted 2014-09-08; First posted 2014-09-18 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; First Relapse
Keywords: Myeloma; Multiple Myeloma; Relapse; Refractory; PCD; IFM/DFCI 2009; Transplantation; Autologous; Pomalidomide; Immunoglobulin; Ig; Free light Chain
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previous IFM/DFCI 2009 arm A (Other): Patients previously randomized into IFM/DFCI 2009 trial arm A (or if transplantation was not done) will receive:
  * The treatment phase:
    * 4 cycles of PCD (Pomalidomide-Cyclophosphamide-Dexamethasone)
  * The consolidation phase:
    * Melphalan 200mg/m2 followed by ASCT (Autologous Stem Cell Transplantation)
    * 2 cycles of PCD (Pomalidomide-Cyclophosphamide-Dexamethasone)
  * The maintenance phase: Until progression or discontinuation for any other reason
    * Pomalidomide and Dexamethasone
  Interventions: Drug: PCD
- Previous transplantation IFM/DFCI 2009 arm B (Other): Patients previously randomized into IFM/DFCI 2009 trial arm B (RVD plus Transplant) will receive:
  * The treatment phase:
    * 4 cycles of PCD (Pomalidomide-Cyclophosphamide-Dexamethasone)
  * The consolidation phase:
    * 5 cycles of PCD (Pomalidomide-Cyclophosphamide-Dexamethasone)
  * The maintenance phase: Until progression or discontinuation for any oher reason
    * Pomalidomide and Dexamethasone
  Interventions: Drug: PCD; Procedure: Autologous transplantation (ASCT)

INTERVENTIONS:
Drug: PCD — STUDY TREATMENT PHASE: All patients
  * 4x 28 days cycles of PCD
  [Pomalidomide: 4mg/day oral route on 21 days per cycle]
  [Cyclophosphamide: 300mg/day oral route on days 1, 8, 15, 22 per cycle]
  [Dexamethasone: 40mg/day oral route on days 1, 2, 3, 4 and 15, 16, 17, 18 per cycle]
  CONSOLIDATION PHASE: depends on previous IFM/DFCI 2009's arm:
  Arm A:
  * Melphalan 200mg/m2 followed by Autologous Transplantation
  * 2x 28 days cycles of PCD, three months post transplantation
  Arm B:
  * 5x 28 days cycles of PCD
  [Pomalidomide: 4mg/day oral route on 21 days per cycle]
  [Cyclophosphamide: 300mg/day oral route on days 1, 8, 15, 22 per cycle]
  [Dexamethasone: 40mg/day oral route on days 1, 8, 15, 22 per cycle]
  MAINTENANCE PHASE: All patients
  - Until progression/relapse or discontinuation for any other reason
  [Pomalidomide: 4mg/day oral route on 21 days per cycle]
  [Dexamethasone: 20mg/day oral route on days 1, 8, 15, 22 per cycle]
  Other Names: Pomalidomide-Cyclophosphamide-Dexamethasone association
Procedure: Autologous transplantation (ASCT) — Arm A:
  •Melphalan 200mg/m2 followed by Autologous Transplantation
  Arms: Previous transplantation IFM/DFCI 2009 arm B

SUMMARY:
Imnovid in combination with dexamethasone is indicated in the treatment of adult patients with relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both lenalidomide (Revlimid) and bortezomib (Velcade), and have demonstrated disease progression on the last therapy.

Patients with relapsed and refractory multiple myeloma who have received bortezomib, lenalidomide, dexamethasone combination, considered to be the multiple myeloma optimal treatment, can access to pomalidomide under marketing authorization only as from third line of treatment.

In France this combination is not authorized for marketing for a first line treatment and only patient randomized in the IFM/DFCI 2009 trial received it.

This study concerns patients previously randomized in the IFM/DFCI 2009 trial who have received bortezomib, lenalidomide and Dexamethasone combination in first line, which at progression/relapse time therapeutic opportunities remained limited and who cannot access pomalidomide under marketing authorization.

This study is a multicentre, phase 2, open label, study testing the triple combination of pomalidomide and cyclophosphamide and dexamethasone (PCD) in multiple myeloma patients who are refractory or in first progression/relapse after a first line treatment with bortezomib and lenalidomide, an IMiDs (an Immuno Modulatory Drug and a proteasome inhibitor) according to the IFM/DFCI 2009 trial.

In the IFM/DFCI trial, patients in arm A received eight cycles of the Velcade-Revlimid-Dexamethasone combination followed by 1 year of lenalidomide maintenance, patients in arm B received 3 cycles of Velcade-Revlimid-Dexamethasone combination plus melphalan 200mg/m2 with an autologous transplantation followed by 2 cycles of Velcade-Revlimid-Dexamethasone combination consolidation and 1 year of lenalidomide maintenance.

This study will contain 3 treatment phases:

* Study treatment phase:

All patients will receive 4 cycles (28 days) of pomalidomide-cyclophosphamide-dexamethasone combination.

* Consolidation phase (depends on the initial randomization in the IFM/DFCI 2009 trial):

  * For patients previously randomized in IFM/DFCI 2009's arm A:

    * Melphalan 200 mg/m2 followed by Autologous Transplantation
    * Three months after, 2 cycles of pomalidomide-cyclophosphamide-dexamethasone combination
  * For patients previously randomized in IFM/DFCI 2009's arm B:

    * 5 cycles of pomalidomide-cyclophosphamide-dexamethasone combination
* Maintenance phase (identical to all patients) subsequent cycles of pomalidomide and Dexamethasone until progression / relapse or discontinuation for any other reason.

For arm B patients, in case relapse occurs at least 12 months after the end of the maintenance IFM/DFCI 2009 trial, they could proceed to a second autologous transplantation and therefore follow the arm A procedure. The decision to proceed to a second transplant will be made by the physician and the patient.

In order to have the same amount of patients enrolled in this trial in the initial Arm A and Arm B of the IFM/DFCI 2009 trial, once 50 patients have been included in either arm A or B, subsequent patients will be eligible if they have not been initially treated as the first 50 patients from either arm.

The primary endpoint is the response rate (Partial Response (PR) or better) after 4 cycles of the triple combination pomalidomide and cyclophosphamide and dexamethasone (PCD) in the studied population using International Myeloma Working Group (IMWG) response criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have been treated in first line within the IFM/DFCI 2009 trial to be treated within the PCD trial in second line
2. Must be able to understand and voluntarily sign an informed consent form
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. Age: 18-70 years
5. Life expectancy >6 months
6. Patients must have progressive (+/- symptomatic) Myeloma as defined by the IMWG criteria with increase of ≥25% from lowest response value in any one or more of the following:

   * Serum M-component and/or (the absolute increase must be ≥0.5 g/dl)
   * Urine M-component and/or (the absolute increase must be ≥200 mg/24h)
   * Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dl
   * Bone marrow plasma cell percentage; the absolute percentage must be ≥10%
   * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
   * Development of hypercalcaemia (corrected serum calcium >11.5 mg/dl or 2.65mmol/l) that can be attributed solely to the plasma cell proliferative disorder.
7. Patients must have a clearly detectable and quantifiable monoclonal M-component value:

   * IgG (serum M-component >10g/l)
   * IgA (serum M-component >5g/l)
   * IgD (serum M-component >0.5g/l)
   * Light chain (serum M-component >1g/l or Bence Jones >200mg/24h)
   * In patients without measurable serum and urine M-protein levels and in the absence of renal failure: when the absolute serum FreeLightChain (sFLC) is ≥100mg/l and an abnormal sFLC K/λ ratio (<0.26 or>1.65) is found.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
9. Adequate bone marrow function, documented within 96 hours prior to treatment without transfusion or growth factor support, defined as:

   * Absolute neutrophils ≥1000/mm3
   * Platelets ≥75000/mm3
   * Hemoglobin ≥8.5g/dl
10. Adequate organ function, documented within 96 hours prior to treatment, defined as:

    * Serum SGOT/AST or SGPT/ALT <3.0 X Upper Limit of Normal (ULN)
    * Serum creatinine clearance (Cockcroft-Gault formula) ≥50 ml/min
    * Serum total bilirubin <2.0 mg/dl
11. Wash out period of at least 2 weeks from previous antitumor therapy or any investigational treatment.
12. Able to take antithrombotic medicines such as low molecular weight heparin or aspirin.
13. Subjects affiliated with an appropriate social security system
14. Agree to abstain from donating blood while taking study drug therapy and for at least 28 days following discontinuation of study drug therapy
15. Agree not to share study medication with another person and to return all unused study drug to the investigator
16. Female subjects of childbearing potential (*) must:

    * Understand the potential teratogenic risk to the unborn child
    * Understand the need and agree to use, and be able to comply with, two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study:

      1. for at least 28 days before starting study drug;
      2. while participating in the study;
      3. dose interruptions; and
      4. for at least 28 days after study treatment discontinuation.

    The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. Females of childbearing potential must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:
    * Highly effective methods:

      * Intrauterine device (IUD)
      * Hormonal (birth control pills, injections, implants)
      * Tubal ligation
      * Partner's vasectomy
    * Additional effective methods:

      * Male condom
      * Diaphragm
      * Cervical Cap

    Because of the increased risk of venous thromboembolism in patients with multiple myeloma taking pomalidomide and cyclophosphamide and dexamethasone, combined oral contraceptive pills are not recommended. If a female subject is currently using combined oral contraception the patient should switch to another one of the highly effective methods listed above. The risk of venous thromboembolism continues for 4-6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.

    Implants and levonorgestrel-releasing intrauterine devices are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia.

    o Agree to have pregnancy testing based on the frequency outlined below.

    Medically supervised pregnancy tests with a minimum sensitivity of 25 mIU/ml must be performed for females of childbearing potential, including females of childbearing potential who commit to complete abstinence:
    * Before starting study drug: females of childbearing potential must have two negative pregnancy tests prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The patient may not receive study drug until the study doctor has verified that the results of these pregnancy tests are negative.
    * During study participation and for 28 days following study drug discontinuation:

    Females of childbearing potential with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following study drug discontinuation.

    If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following study drug discontinuation.

    *Criteria for women of childbearing potential: This protocol defines a female of childbearing potential as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
17. Male subjects must:

    * Practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
    * Agree not to donate semen or sperm during study drug therapy and for at least 28 days following discontinuation of study drug.

Exclusion Criteria:

1. Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation
2. Primary amyloidosis or myeloma complicated by amyloidosis
3. Pregnant or breast feeding females
4. Use of any other experimental drug or therapy within 2 weeks before study treatment initiation (except local radiotherapy and/or corticosteroid until dose of dexamethasone 160mg)
5. Known positive for HIV or Active infectious hepatitis, type B or C
6. Patients with non-secretory MM
7. Prior history of malignancies within 10 years
8. Evidence of Central Nervous System (CNS) involvement
9. Any >grade 2 toxicity unresolved
10. Peripheral neuropathy >grade 2
11. Known hypersensitivity to thalidomide, lenalidomide, cyclophosphamide or dexamethasone
12. Ongoing active infection, especially ongoing pneumonitis
13. Participant with clinical signs of heart or coronary failure, or evidence of Left Ventricular Ejection Fraction (LVEF) inferior to 40%.

    Participant with myocardial infarction within 6 months prior to enrolment or have New York Heart Association (NYHA) Class III or IV heart failure, and controlled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
14. Inability or unwillingness to comply with birth control requirements
15. Unable to take antithrombotic medicines at study entry
16. Unable to take corticotherapy at study entry
17. Scheduled vaccination with a live agent such as yellow fever vaccine
18. Individually deprived of liberty or placed under the authority of a tutor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Response rate (Partial response (PR) or better) | 4 months after treatment initiation
  after 4 cycles of the triple association

SECONDARY OUTCOMES:
Safety : incidence of Adverse Events and Serious Adverse Events and laboratory abnormalities | from consent to 28 days after the last dose
  using National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTC AE) V4.03

OTHER OUTCOMES:
Time to response and response duration | every 28 days until progression/relapse or discontinuation
  Time to response (from the date of inclusion to the date of the first observation of response) and response duration (time between first documentation of response and disease progression).
Time to Disease Progression | every 28 days until progression/relapse or discontinuation
  from first dose to first observation of disease progression
Overall Survival (OS) | 5 years from last study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: KUHNOWSKI Frederique, MD, Principal Investigator — Institut Curie
Locations (30):
- France (30):
  - CHRU Hopital Sud, Amiens
  - Centre Hospitalier de la côte Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - ICH - Hôpital A. Morvan, Brest
  - Institut d'Hématologie de Basse Normandie - IHBN, Caen
  - Chu Estaing, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Centre Hospitalier Général, Dunkirk
  - Chru Grenoble, Grenoble
  - Centre Hospitalier départemental de Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHRU - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Institut Paoli Calmette, Marseille
  - Hopital Emile Muller, Mulhouse
  - CHU de Nantes, Nantes
  - CHU Carémeau, Nîmes
  - Institut Curie, Paris
  - CHRU Hopital Saint Antoine, Paris
  - CHRU Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHRU Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Institut Universitaire du Cancer Toulouse-Oncopôle (IUCT-O), Toulouse
  - CHRU Hopital Bretonneau, Tours
  - CHRU Hopitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garderet L, Kuhnowski F, Berge B, Roussel M, Devlamynck L, Petillon MO, Escoffre-Barbe M, Lafon I, Facon T, Leleu X, Karlin L, Perrot A, Stoppa AM, Royer B, Chaleteix C, Tiab M, Araujo C, Lenain P, Macro M, Belhadj K, Ikhlef S, Hulin C, Loiseau HA, Attal M, Moreau P. Pomalidomide and dexamethasone until progression after first salvage therapy in multiple myeloma. Br J Haematol. 2023 Jun;201(6):1103-1115. doi: 10.1111/bjh.18772. Epub 2023 Mar 27. PMID 36974007
- [Derived] Garderet L, Kuhnowski F, Berge B, Roussel M, Escoffre-Barbe M, Lafon I, Facon T, Leleu X, Karlin L, Perrot A, Moreau P, Marit G, Stoppa AM, Royer B, Chaleteix C, Tiab M, Araujo C, Lenain P, Macro M, Voog E, Benboubker L, Allangba O, Jourdan E, Orsini-Piocelle F, Brechignac S, Eveillard JR, Belhadj K, Wetterwald M, Pegourie B, Jaccard A, Eisenmann JC, Glaisner S, Mohty M, Hulin C, Loiseau HA, Mathiot C, Attal M. Pomalidomide, cyclophosphamide, and dexamethasone for relapsed multiple myeloma. Blood. 2018 Dec 13;132(24):2555-2563. doi: 10.1182/blood-2018-07-863829. Epub 2018 Oct 3. PMID 30282798